CLINICAL TRIAL: NCT05567107
Title: The Effect of Foot Massage After Open Heart Surgery on Postoperative Pain, Sleep Quality and Mood of Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Beyzanur Kızıloğlu, PhD student, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BKiziloglu
Record Dates: First submitted 2022-09-22; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Pain, Postoperative; Sleep Disturbance; Mood; Bypass Complication
Keywords: sleep quality; open heart surgery; foot massage; pain; mood
MeSH Terms: conditions — Pain, Postoperative; Parasomnias; Sleep Initiation and Maintenance Disorders; Pain | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group: applied foot massage (Experimental): Scales were applied preoperative to the patients. After being discharged from the intensive care unit in the postoperative period, the scales were applied without any intervention on the first day of hospitalization (day 0). Pain intensity was evaluated according to the Visual Comparison Pain Scale and classical foot massage was applied to patients who stated that they had 4 or more pain. After leaving the intensive care unit in the postoperative period, the scales were applied on the 2nd day (day 1) when the patient came to the service. After the scales, foot massage was applied again. After leaving the intensive care unit in the postoperative period, the scales were applied on the third day (day 2) when the patient came to the service. After the scales, foot massage was applied again. After the patient was discharged from the intensive care unit in the postoperative period, the scales were applied on the fourth day (3rd day) when they came to the service.
  Interventions: Other: massage
- control group: unapplied foot massage (No Intervention): Each data collection tool was collected without applying foot massage, as in the experimental group patients. While the patients in the control group received only analgesic treatment postoperatively, the patients in the experimental group received foot massage in addition to the analgesic treatment. Only routine nursing care was given to the patients in the control group postoperatively.

INTERVENTIONS:
Other: massage — Classical foot massage was applied by the researcher with efflorescence, superficial friction and petrissage techniques for 10 minutes on each foot.
  Arms: experimental group: applied foot massage

SUMMARY:
The randomized controlled experimental study was conducted in the cardiovascular surgery clinic of Atatürk University Health Practice and Research Center between April 2021 and September 2021.The research sample consisted of 91 patients who met the research criteria. Since exclusion criteria were met in 15 patients during the research process, the study was completed with 76 patients. Descriptive Information Form, Visual Analog Scale, State-Trait Anxiety Scale, Visual Analog Sleep Scale and Hospital Anxiety and Depression Scale were used as data collection tools. All scales were applied to the patients preoperatively. According to the Postoperative Visual Analog Scale, the patients in the experimental group who stated that they had more than 4 pains were given foot massage for a total of 20 minutes, 10 minutes on each foot. After the surgery, classical foot massage was applied to the patients for 3 consecutive days, including the day they came to the service from the intensive care unit. One day after each application, the patients' pain, sleep quality and mood levels were examined. Data were collected by applying the same procedure steps without foot massage to the patients in the control group.

DETAILED DESCRIPTION:
Pain still remains a major problem in patients undergoing coronary artery bypass graft surgery. Pain and anxiety are conditions that should be evaluated together and affect each other. Anxiety has a significant effect on the reduction or increase in post-operative pain. Pain experienced after surgery increases the anxiety of the individual. Increasing anxiety level negatively affects sleep quality. The inability to manage the pain experienced in the early postoperative period and the associated anxiety negatively affect the healing process, increasing the risk of complications that may occur after the surgery, which negatively affects the quality of life. It also increases mortality and morbidity rates. Pain management is very important because of the negative effects seen due to pain. It is seen that there are many pharmacological and non-pharmacological methods used to prevent pain and anxiety experienced after surgical intervention. One of these methods is massage, which is known for its therapeutic and healing effects and has a positive effect on the body. It is predicted that with the foot massage applied after coronary artery bypass graft surgery, the postoperative pain and anxiety level of the patients will decrease, it will have a positive effect on their mood and their sleep quality will increase. In addition, it is thought that with the increase of studies on the application of foot massage in patients who have undergone coronary artery bypass graft surgery, a non-pharmacological routine application can be created on patients in surgical services and the level of satisfaction in nursing can be increased.

ELIGIBILITY:
Inclusion Criteria:

* Those who agree to participate in the research
* Those who have planned coronary artery bypass graft surgery between the specified dates
* 18 years of age or older
* Not having visual/verbal/auditory communication difficulties and mental disabilities that would prevent him/her from expressing the explained information correctly.
* Hypertension under control
* Those who state that they have 4 or more post-operative GCS pain
* For patients in the experimental group; infectious disease of the foot skin, local infection, open lesion/wound, scar tissue, edema, hematoma, thrombophlebitis, deep vein thrombosis, coagulation disorder, varicose veins, osteoporosis, osteomyelitis, hepatitis, inflammatory and degenerative joint diseases, diabetes-induced neuropathy, toes patients without deformities, recent fractures, dislocations, ruptures of muscle fibers, tendons, or fascia

Exclusion Criteria:

◾Patients who develop any complications after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | [Time Frame: up to 24 hours]
  The visual analog scale was used to evaluate the pain severity of the patient. It is a self-reported scale in the form of a 10-cm ruler indicating no pain at one end and unbearable pain at the other. Accordingly, the patient is told to evaluate his/her pain between 0 and 10, with 0 cm indicating "no pain" and 10 cm indicating "unbearable pain"
State-Trait Anxiety İnventory (STAI-I, STAI-II) | [Time Frame: up to 24 hours]
  It is a test developed by Spielberger et al. that measures state and trait anxiety levels. Its validity and reliability in Turkey was done by O#ner and Le Compte. The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
Visual Comparison Sleep Scale | [Time Frame: up to 24 hours]
  Scoring in this scale, whose Turkish version consists of 10 items, was formed by reversing the 2nd, 4th, 8th and 9th statements. Each item in the scale was evaluated by visual comparison technique by showing it on the chart between 0 (on the left end) and 100 (on the right end). The score obtained from the scale is between 0-1000. An increase in the score obtained from the scale indicates a decrease in sleep quality.
Hospital Anxiety and Depression Scale | [Time Frame: up to 24 hours]
  It consists of two subscales, depression and anxiety. Each subscale includes 7 items. There are 14 items in total. While summing the scores of items 1, 3, 5, 7, 9, 11 and 13 for the Anxiety Subscale of the Hospital Anxiety and Depression Scale; For the Depression Sub-Scale, the scores of items 2, 4, 6, 8, 10, 12 and 14 are added. Items 3, 5, 6, 8, 10, 11, and 13 of the Anxiety Sub-Scale of the Hospital Anxiety and Depression Scale show gradually decreasing severity and are scored in a 4-point Likert scale as 3, 2, 1, 0. Items 2, 4, 7, 9, 12 and 14 of the Depression Subscale of the Hospital Anxiety and Depression Scale show increasing severity and are scored as 0, 1, 2, 3 on a 4-point Likert scale. The lowest score that patients can get from the Anxiety and Depression Subscales is 0, and the highest score is 21.

CONTACTS AND LOCATIONS:
Locations (1):
- Beyzanur Kızıloğlu, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No